CLINICAL TRIAL: NCT02992392
Title: Comparison of the Clinical Effects of Two Tear Substitutes in Patients With Dry Eye Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xingwu Zhong, MD PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-007
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Dry Eye
Keywords: Tear film; Lipid layer; Liposic; Tears Naturale Forte
MeSH Terms: conditions — Dry Eye Syndromes | interventions — carbomer; Dextrans

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposic (Experimental): Liposic was applied to one eye of patients in this group
  Interventions: Drug: Liposic
- Tears Naturale Forte (Experimental): Tears Naturale Forte was applied to one eye of patients in this group
  Interventions: Drug: Tears Naturale Forte

INTERVENTIONS:
Drug: Liposic — one eye of the participant recieved Lipoic
  Other Names: Carbomer
  Arms: Liposic
Drug: Tears Naturale Forte — the other eye of the participant recieved Tears Naturale Forte
  Other Names: DEXTRAN/HYPROMELLOSE/GLYCERIN
  Arms: Tears Naturale Forte

SUMMARY:
With the potential to address evaporative dry eye, Liposic and Tears Naturale Forte have been developed in which phospholipid liposomes are delivered to the tear film via the surface of the closed eyelid. This study compare the effects of Liposic and Tears Naturale Forte application on the lipid and stability of the tear film in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 20 years(range from 20 year to 25 years)
* The value of OSDI is over 12
* NBUT is less 5 seconds
* Schirmer 1 test is less 10mm
* The basical lipid layer grade is 1-2

Exclusion Criteria:

* Any corneal,conjunctival, or eyelid abnormalities; conjunctivitis; current ocular infection; photophobia that may cause reflex tearing or difficulty in evaluating the patient's lipid layer;
* Known allergic sensitivity to any of the ingredients in Liposic or Tears Naturale Forte

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
scale of Schirmer I test | up to 3 months after tear substitutes apply
scale of corneal fluorescein staining | up to 3 months after tear substitutes apply
scale of noninvasive tear breakup time | up to 3 months after tear substitutes apply
scale of tear meniscus height | up to 3 months after tear substitutes apply
lipid layer grade | up to 3 months after tear substitutes apply
questionnaire of ocular surface disease index | up to 3 months after tear substitutes apply

SECONDARY OUTCOMES:
subjective comfort | up to 3 months after tear substitutes apply
  Subjective comfort was established at each time-point by asking subjects, firstly, to relate their comfort to baseline in each eye (more comfortable/no different/less comfortable) . secondly, to express a preference for their more comfortable eye (right eye/left eye/no difference)

CONTACTS AND LOCATIONS:
Overall Officials: Xingwu Zhong, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Hainan Eye Hospital, Zhongshan Ophthalmic Center of Sun Yat-sen University, Haikou, Hainan, China